CLINICAL TRIAL: NCT03528928
Title: Evaluation of Pelvic Floor Muscle With Surface Electrical Stimulation
Brief Title: Viewing Surface Electrical Stimulation on Pelvic Floor With Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elidah, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 0318
Record Dates: First submitted 2018-05-07; First posted 2018-05-18 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Floor Disorders
Keywords: pelvic floor; electrical stimulation; bladder; ultrasound
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: Surface electrical stimulation, Elitone by Elidah, Inc.
Masking Description: The patient was not allowed to see the ultrasound screen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Surface electrical stimulation (Experimental): Each subject did a Kegel pelvic floor contraction, had the surface electrical stimulation turned on at highest comfortable intensity, did a Kegel contraction with surface electrical stimulation on, and had second electrical stimulation turned on.
  Interventions: Device: Surface electrical stimulation

INTERVENTIONS:
Device: Surface electrical stimulation — Thin electrode with four conductive areas placed over the perineal area.
  Other Names: Elitone

SUMMARY:
Subjects will place a surface electrode on their perineal area after a bladder-filling protocol. Transabdominal ultrasound will image the base of the bladder at rest, voluntary pelvic floor contraction, with the surface electrical stimulation and with a combined pelvic floor contraction and electrical stimulation active.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-80y
* Gender: female

Exclusion Criteria:

* Moderate-severe stress incontinence*: As determined by self-reported >3 accidents in 24-hr period
* Currently pregnant, may be pregnant (Unsure pre and peri-menopausal women should take a pregnancy test.)
* Active urinary tract infection (UTI)
* Pelvic pain, Painful bladder syndrome, underlying neurologic/neuromuscular disorder that may impact ability to partake in the trial
* implanted cardiac device or untreated cardiac arrhythmia
* Obesity as defined by BMI >= 30 (height, weight recorded)
* Anyone with impaired decision making, drug or alcohol dependence, or potentially suicidal.
* Anyone who lacks the capacity to consent for themselves or who requires a legal representative to give informed consent * Stress urinary incontinence: as determined by an answer of "Yes" to a standard question (from King's Health Questionnaire): "Do you lose urine with physical activities such as coughing, sneezing, running?"

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2018-04-17 (Actual); Study Completion 2019-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wome's Health Advantage, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Surface Electrical Stimulation
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Surface Electrical Stimulation
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
BMI [Mean (Standard Deviation); unit: lbs/ in^2] | 24.9 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Movement of the Bladder
Description: Visualization of movement of the bladder with use of device by transabdominal ultrasound was captured and the measurement is measured in pixels for centroid magnitude displacement.
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: pixels
Arm/Group | Surface Electrical Stimulation
Number analyzed (Participants) | 8
pixels | 23.1 (11.7)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Same as clinical trials definition
Arm/Group | Surface Electrical Stimulation
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT03528928/Prot_SAP_001.pdf